CLINICAL TRIAL: NCT06314854
Title: The Effect of Running Water Sound Listened to Patients During Hemodialysis on Invasive Pain and Anxiety Experienced During Cannulation
Brief Title: The Effect of Running Water Sound Listened to Patients During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Aylin Aydin Sayilan, Principal Investigator, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P202300046
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hemodialysis Patients
Keywords: anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): During the cannulation process, the experimental group will listen to the sound of flowing water throughout the process through the researcher's smartphone. The experimental and control groups will be administered VAS before, during and after each cannulation, and the State and Trait Anxiety Scale will be administered before the dialysis session and after the 12th first session.
  Interventions: Other: Running water sound
- Control Group (No Intervention): The control group will be provided with standard care and no intervention will be made. A total of 12 sessions will be followed in both groups.

INTERVENTIONS:
Other: Running water sound — Running water sound for experimental group Standard care for control group
  Arms: Experimental Group

SUMMARY:
It is known that being in nature and the visual perception of nature positively affects an individual's mood and self-confidence. Studies have reported that natural sounds have a positive effect in situations such as pain, anxiety, and stress. This finding means that listening to natural sounds may be a simple and easily accessible intervention that can positively impact key human stress systems.

Although many non-pharmacological methods are used in the literature to reduce the invasive pain and anxiety experienced by hemodialysis (HD) patients during cannulation, the most popular recently; However, we aimed to determine the effect of the sound of running water, which we have not yet encountered in dialysis patients, on invasive pain and anxiety experienced during fistula access.

DETAILED DESCRIPTION:
In this study; Between 15 December 2023 and 15 March 2024, patients receiving dialysis will be included in the Dialysis Service of two hospitals in western of Turkey which havedialysis for 3 days a week.

The sample calculation was determined using power analysis based on a previous study. (Çetinkaya, Karabulut (2010). The sample size of the study was calculated as at least 30 patients, for each group that met the sampling criteria. The population of the research was determined as 74 people. The number of patients who met the inclusion criteria was 68, and these patients were assigned to the experimental (34 patients) and control (34 patients) groups by an independent statistician with the help of a computer program (randomizer.org).

Patients over the age of 18, who are volunteers, who undergo dialysis 3 days a week, who do not have any communication problems and who do not use any psychiatric medication will be included in the study. Patients who do not meet the inclusion criteria will be excluded from the study.

Dialysis sessions are held 3 days a week, between 08.00-16.00, on Mon-Wed-Fri and Tuesday-Thurs-Sat.

All patients who volunteer to participate in the study will be included in the study. During the cannulation process, the experimental group will listen to the sound of flowing water throughout the process with the help of the researcher's smartphone. VAS scale will be applied to the experimental and control groups after each cannulation, and the State and Trait Anxiety Scale will be applied before the first dialysis session and after the 12th session. The control group will receive standard care. A total of 12 sessions will be followed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* between 18 - 65 years
* not have communication problem
* Patients receiving dialysis 3 days a week
* Have cannulation

Exclusion Criteria:

* under 18- over 65 years
* Have communication problems
* Not have dialysis 3 days a week
* Have not cannulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | nearly 40 days
  VAS

SECONDARY OUTCOMES:
State and Trait Anxiety Assessment | nearly 40 days
  STAI I AND STAI II

CONTACTS AND LOCATIONS:
Locations (1):
- Aas, Kırklareli, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided